CLINICAL TRIAL: NCT00551018
Title: Efficacy and Safety of VICRIVIROC in HIV-Infected Treatment-Naïve Subjects
Brief Title: Efficacy and Safety of VICRIVIROC in HIV-Infected Treatment-Naïve Subjects (Study P04875)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04875
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — vicriviroc; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Racivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vicriviroc + Reyataz + ritonavir (Experimental): vicriviroc 30 mg tablet QD + Reyataz® (atazanavir sulfate) 300 mg (1x300 mg capsule or 2x150 mg capsules) QD + Norvir® (ritonavir) 100 mg capsule QD
  Interventions: Drug: Vicriviroc
- Truvada® + Reyataz + ritonavir (Active Comparator): Truvada® 200/300 combination tablet QD + Reyataz® (atazanavir sulfate) 300 mg (1x300 mg capsule or 2x150 mg capsules) QD + Norvir® (ritonavir) 100 mg capsule QD
  Interventions: Drug: emtricitabine and tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: Vicriviroc — one 30 mg tablet QD
  Other Names: SCH 417690; VCV
  Arms: Vicriviroc + Reyataz + ritonavir
Drug: emtricitabine and tenofovir disoproxil fumarate — one 200/300 combination tablet QD
  Other Names: Truvada®, a combination of Emtriva® (emtricitabine 200 mg) and Viread® (tenofovir disoproxil fumarate 300 mg); emtricitabine + tenofovir DF; FTC + TDF
  Arms: Truvada® + Reyataz + ritonavir

SUMMARY:
Vicriviroc (vye-kri-VYE-rock) is an investigational drug (not yet approved by Government Regulatory Authorities for commercial use) that belongs to a new class of drugs, called CCR5 receptor blockers. This group of drugs blocks one of the ways HIV enters T-cells (the cells that fight infection). Previous smaller studies in HIV treatment-experienced patients, have shown that vicriviroc is safe and effective. The purpose of this study is to evaluate the virologic efficacy of vicriviroc combined with ritonavir-boosted Reyataz® in HIV-infected treatment-naïve subjects.

DETAILED DESCRIPTION:
This is a randomized, open-label, active-controlled, parallel-group, multi-center study of vicriviroc maleate in treatment-naïve subjects infected with CCR5-tropic HIV. The study will compare the virologic benefit of vicriviroc combined with ritonavir-boosted Reyataz to a control group receiving Truvada plus ritonavir-boosted Reyataz. Interim analyses will be performed when the first cohort of 80 subjects have completed 24 weeks and 48 weeks of treatment. The second cohort of 120 subjects will be enrolled after the first interim analysis; a third interim analysis will be performed when subjects in this second cohort have completed 24 weeks of treatment. The primary efficacy analysis will be conducted when all 200 subjects from both stages have completed 48 weeks of treatment or discontinued. The final analysis will be performed at Week 96, when all 200 subjects have completed 96 weeks of treatment or discontinued. If vicriviroc is shown to provide benefit at the studied dose, study participants in the vicriviroc arm who complete 96 weeks of treatment may continue in a protocol extension, where they will be offered vicriviroc free of charge until the drug is commercially available in their location or until the sponsor terminates the clinical development of vicriviroc.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects at least 18 years old or minimum age that defines an adult as determined by local regulatory authorities or legal requirements) of either sex or any race with CCR5-tropic HIV infection.
* Cumulative lifetime anti-retroviral therapy exposure of at most 4 weeks (with the exception of prophylaxis to prevent mother-to-child transmission, and in this case, if no antiretroviral resistance is expected to have developed) and none in the 8 weeks preceding randomization.
* A CD4 cell count of at least 100 cells/(cubic mm) at Screening (or as specified by local treatment guidelines).
* HIV ribonucleic acid (RNA) must be at least 2000 copies/mL at Screening.
* Subjects should meet International AIDS Society (IAS), Department of Health and Human Services (DHSS), or local recommendations for initiation of antiretroviral therapy (ART).
* Platelet count must be at least 50,000/microL, hemoglobin at least 8 g/dL, absolute neutrophil count at least 1000/microL, serum creatinine <2.0 mg/dL (154 micromol/L), and SGOT/SGPT (serum glutamic oxaloacetic transaminase/serum glutamic pyruvic transaminase) at most 3 x upper limit of normal at Screening. Other clinical laboratory tests must be within normal limits or clinically acceptable to the investigator.
* Female subjects of childbearing potential must be using a medically accepted method of birth control prior to Screening and agree to continue its use during the study, or must have been surgically sterilized.
* Female subjects of childbearing potential must have a negative serum beta-hCG (human chorionic gonadotropin) pregnancy test at Screening and a negative urine beta-hCG pregnancy test on Day 1 prior to dosing.

Exclusion Criteria:

* Female subjects of childbearing potential who are breastfeeding, pregnant, or planning to become pregnant.
* Subjects with intercurrent illness, vaccinations, or who have used immunomodulators (within the 4 week period prior to randomization) that could influence plasma HIV RNA levels.
* CXCR4 or dual-mixed (CXCR4 and CCR5) tropism.
* Subjects with primary resistance mutations to any of proposed components of the study arms.
* Subjects with active opportunistic infection or malignancy.
* Subjects with seizure disorder requiring ongoing anti-seizure therapy or with a history of a seizure disorder who are, in the judgment of the investigator, at risk for seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2007-12; Primary Completion 2010-05 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in log10 HIV RNA | Week 48

SECONDARY OUTCOMES:
Proportion of subjects with plasma HIV RNA <50 copies/mL | Week 48